CLINICAL TRIAL: NCT02139306
Title: A Phase 3 Efficacy and Safety Study of Ataluren (PTC124®) in Patients With Nonsense Mutation Cystic Fibrosis
Brief Title: Study of Ataluren in Nonsense Mutation Cystic Fibrosis (ACT CF)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: PTC Therapeutics (Industry)
Collaborators: Cystic Fibrosis Foundation (Other); ECFS-Clinical Trial Network (ECFS-CTN) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PTC124-GD-021-CF; 2013-004581-34 (EudraCT Number)
Record Dates: First submitted 2014-05-13; First posted 2014-05-15 (Estimated); Results first posted 2020-05-14 (Actual); Last update posted 2020-05-14 (Actual); Status verified 2020-05

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis | interventions — ataluren

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ataluren (PTC124®) (Experimental): Participants received ataluren as oral powder for suspension at the dosages of 10, 10, and 20-mg/kg at morning, midday and evening, respectively for 48 weeks of treatment duration or until treatment discontinuation.
  Interventions: Drug: Ataluren (PTC124®)
- Placebo (Placebo Comparator): Participants received matching placebo orally at morning, midday and evening for 48 weeks of treatment duration or until treatment discontinuation.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ataluren (PTC124®) — Oral Ataluren TID
  Arms: Ataluren (PTC124®)
Drug: Placebo — Oral Placebo TID
  Arms: Placebo

SUMMARY:
This is a Phase 3, international, multicenter, randomized, double-blind, placebo-controlled, efficacy and safety study of ataluren in patients with nonsense mutation cystic fibrosis (nmCF) not receiving chronic inhaled aminoglycosides.

DETAILED DESCRIPTION:
This study is to enroll 208 subjects (184 fully evaluable) with nonsense-mutation-mediated CF who are at least 6 years of age and have an forced expiratory volume in 1 second (FEV1) >= 40% and <= 90% of predicted. Subjects will be stratified based on age, inhaled antibiotic use, and baseline FEV1, and will be randomized in a 1:1 ratio to receive oral ataluren administered 3 times per day (TID) at respective morning, midday, and evening doses of 10-, 10-, and 20-mg/kg or placebo. Based on the results of a previously conducted study, patients treated with chronic inhaled aminoglycosides (including TOBI) will not be eligible for participation. Spirometry measurement at the screening visit will establish patient eligibility for inclusion based on lung function. FEV1 stability will be assessed during the approximately 4-week screening period, at the conclusion of which patients will be required to demonstrate a relative change in %-predicted FEV1 of less than 15% when compared to the screening value. Assessments will be performed every 8 weeks, depending upon the outcome measure.

ELIGIBILITY:
Inclusion Criteria:

* Evidence of signed and dated informed consent/assent document(s) indicating that the subject (and/or his parent/legal guardian) has been informed of all pertinent aspects of the trial
* Age >=6 years.
* Body weight >=16 kg.
* Sweat chloride >60 milliequivalent per liter (mEq/L)
* Documentation of the presence of a nonsense mutation in at least 1 allele of the cystic fibrosis transmembrane conductance regulator (CFTR) gene, as determined by genotyping performed at a laboratory certified by the College of American Pathologists (CAP), or under the Clinical Laboratory Improvement Act/Amendment (CLIA), or by an equivalent organization
* Verification that a blood sample has been drawn for sequencing of the CFTR gene
* Ability to perform a valid, reproducible spirometry test using the study-specific spirometer with demonstration of an FEV1 >=40% and <=90% of predicted
* Demonstration at Visit 2 of a valid %-predicted FEV1 within 15% of the Screening % predicted FEV1 value
* Resting oxygen saturation (as measured by pulse oximetry) >=92% on room air.
* Confirmed screening laboratory values within pre-specified ranges
* In subjects who are sexually active, willingness to abstain from sexual intercourse or employ a barrier or medical method of contraception during the study drug administration and 60-day follow-up period
* Willingness and ability to comply with all study procedures and assessments, including scheduled visits, drug administration plan, study procedures, laboratory tests, and study restrictions

Exclusion Criteria:

* Known hypersensitivity to any of the ingredients or excipients of the study drug
* Previous participation in the Phase 3 trial of ataluren (PTC124-GD-009-CF).
* Any change (initiation, change in type of drug, dose modification, schedule modification, interruption, discontinuation, or re-initiation) in a chronic treatment/prophylaxis regimen for Cystic Fibrosis (CF) or for CF-related conditions within 4 weeks prior to screening
* Chronic use of inhaled aminoglycosides (eg, tobramycin) or use of inhaled aminoglycosides within 4 weeks prior to screening.
* Exposure to another investigational drug within 4 weeks prior to screening
* Ongoing participation in any other therapeutic clinical trial
* Evidence of pulmonary exacerbation or acute upper or lower respiratory tract infection (including viral illnesses) within 3 weeks prior to screening
* Treatment with intravenous antibiotics within 3 weeks prior to screening
* Ongoing immunosuppressive therapy (other than corticosteroids)
* Ongoing warfarin, phenytoin, or tolbutamide therapy
* History of solid organ or hematological transplantation
* Major complications of lung disease (including massive hemoptysis, pneumothorax, or pleural effusion) within 8 weeks prior to screening
* Known portal hypertension
* Positive hepatitis B surface antigen, hepatitis C antibody test, or human immunodeficiency virus (HIV) test
* Pregnancy or breast-feeding
* Current smoker or a smoking history of >=10 pack-years (number of cigarette packs/day x number of years smoked).
* Prior or ongoing medical condition (eg, concomitant illness, alcoholism, drug abuse, psychiatric condition), medical history, physical findings, electrocardiogram (ECG) findings, or laboratory abnormality that, in the investigator's opinion, could adversely affect the safety of the subject, makes it unlikely that the course of treatment or follow-up would be completed, or could impair the assessment of study results

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 279 (Actual)
Dates: Start 2014-08 (Actual); Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph McIntosh, MD, Study Director — PTC Therapeutics
Locations (88):
- United States (30):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Pulmonary Associates of Mobile PC, Mobile, Alabama
  - Miller Children's Hospital Long Beach, Long Beach, California
  - Children's Hospital Los Angeles, Los Angeles, California
  - Children's Hospital and Research Center at Oakland, Oakland, California
  - Stanford University-Children's Hospital, Palo Alto, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Nemours Children's Clinic, Jacksonville, Florida
  - University of Miami, Miami, Florida
  - Miami Children's Hospital, Miami, Florida
  - All Children's Hospital, St. Petersburg, Florida
  - Ann and Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - Indiana University, Indianapolis, Indiana
  - Children's Hospital Boston, Boston, Massachusetts
  - Washington University, St Louis, Missouri
  - Monmouth Medical Center, Long Branch, New Jersey
  - Morristown Medical Center, Morristown, New Jersey
  - Beth Israel Medical Center, New York, New York
  - New York University Langone Medical Center, New York, New York
  - Columbia University Medical Center, New York, New York
  - SUNY Upstate Medical University, Syracuse, New York
  - University of Cincinnati, Cincinnati, Ohio
  - Rainbow Babies & Children's Hospital, Cleveland, Ohio
  - Santiago Reyes, MD, Oklahoma City, Oklahoma
  - Penn State Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Drexel University College of Medicine, Philadelphia, Pennsylvania
  - Texas Children's Hospital, Houston, Texas
  - University of Texas Health Science Center, Tyler, Texas
  - Childrens Hospital of Wisconsin, Milwaukee, Wisconsin
- Argentina (3):
  - Hospital Universitario Austral, Buenos Aires
  - Hospital de Niños Dr. Ricardo Gutiérrez, Buenos Aires
  - Hospital de Niños Superiora Sor Maria Ludovica, La Plata
- Australia (3):
  - Royal Adelaide Hospital, Adelaide
  - Prince Charles Hospital, Chermside
  - Princess Margaret Hospital, Perth
- Belgium (3):
  - Hôpital Universitaire des Enfants Reine Fabiola, Brussels
  - University Hospital Brussels, Brussels
  - University Hospital Leuven, Leuven
- Brazil (2):
  - Hospital Sao Lucas Da Pontificia Universidade Catolica Do Rio Grande Do Sul, Porto Alegre
  - Instituto da Criança - Hospital das Clínicas, São Paulo
- Bulgaria (2):
  - University Mulitiprofile Hospital for Active Treatment Sveti Georgi EAD, Plovdiv
  - University Multiprofile Hospital for Active Treatment Aleksandrovska EAD, Sofia
- Canada (4):
  - Clinical Research Institute of Montreal, Montreal
  - CHU de Quebec - Hopital CHUL, Québec
  - University of Toronto Hospital for Sick Children, Toronto
  - British Columbia Children's Hospital, Vancouver
- France (5):
  - Hôpital Femme-Mère-Enfant, Bron
  - Hôpital Arnaud de Villeneuve, Montpellier
  - Hôpital Necker-Enfants Malades, Paris
  - Centre de Perharidy, Roscoff
  - Centre Hospitalier Regional Sud Reunion, Saint-Pierre
- Germany (7):
  - Charité Universitätsmedizin Berlin, Berlin
  - St. Josef Hospital GmbH, Bochum
  - Universitätsklinikum Köln, Cologne
  - Christiane Herzog CF-Zentrum, Frankfurt am Main
  - Universitätsklinikum Jena, Jena
  - LMU Klinikum der Universität München, München
  - Dr. Von Haunersches Kinderspital, München
- General Hospital of Thessaloniki Ippokration, Thessaloniki, Greece
- Israel (2):
  - Meyer Children's Hospital, Haifa
  - Hadassah University Hospital, Jerusalem
- Italy (6):
  - Ospedali Riuniti di Ancona, Ancona
  - Azienda Ospedaliera A Meyer, Florence
  - Lombardia Cystic Fibrosis Center, Milan
  - Ospedale Pediatrico Bambino Gesù IRCCS, Roma
  - Azienda Policlinico Umberto I, Rome
  - University of Verona, Verona
- Netherlands (3):
  - Radboud University, Nijmegen
  - Erasmus MC, Rotterdam
  - Hagaziekenhuis, The Hague
- Poland (4):
  - Szpital Dzieciecy Polanki im Macieja Plazynskiego w Gdansku, Gdansk
  - NZOZ Sanatorium Cassia-Villa Medica, Rabka-Zdrój
  - NZOZ Podkarpacki Osrodek Pulmonologii i Alergologii, Rzeszów
  - Instytut Matki I Dziecka, Warsaw
- Spain (6):
  - Hospital Universitario Vall d'Hebron, Barcelona
  - Hospital University, Barcelona
  - Hospital Sant Joan de Deu, Esplugues de Llobregat
  - Hospital Regional Universitario de Malaga, Málaga
  - Hospital de Sabadell, Consorci Sanitari Parc Tauli, Sabadell
  - Hospital Universitario Virgen del Rocio, Seville
- United Kingdom (7):
  - Birmingham Children's Hospital NHS Foundation Trust, Birmingham
  - Heart of England NHS Foundation Trust, Birmingham
  - Southern General Hospital, Glasgow
  - St James's University Hospital, Leeds
  - Royal Brompton Hospital, London
  - Llandough Hospital, Penarth
  - Southampton University Hospitals NHS Trust, Southampton

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Aslam AA, Sinha IP, Southern KW. Ataluren and similar compounds (specific therapies for premature termination codon class I mutations) for cystic fibrosis. Cochrane Database Syst Rev. 2023 Mar 3;3(3):CD012040. doi: 10.1002/14651858.CD012040.pub3. PMID 36866921
- [Derived] VanDevanter DR, Hamblett NM, Simon N, McIntosh J, Konstan MW. Evaluating assumptions of definition-based pulmonary exacerbation endpoints in cystic fibrosis clinical trials. J Cyst Fibros. 2021 Jan;20(1):39-45. doi: 10.1016/j.jcf.2020.07.008. Epub 2020 Jul 15. PMID 32682670
- [Derived] Konstan MW, VanDevanter DR, Rowe SM, Wilschanski M, Kerem E, Sermet-Gaudelus I, DiMango E, Melotti P, McIntosh J, De Boeck K; ACT CF Study Group. Efficacy and safety of ataluren in patients with nonsense-mutation cystic fibrosis not receiving chronic inhaled aminoglycosides: The international, randomized, double-blind, placebo-controlled Ataluren Confirmatory Trial in Cystic Fibrosis (ACT CF). J Cyst Fibros. 2020 Jul;19(4):595-601. doi: 10.1016/j.jcf.2020.01.007. Epub 2020 Jan 23. PMID 31983658
- See also: Related Info — http://www.ptcbio.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted from 15 August 2014 to 02 November 2016.
Groups:
- Ataluren: Participants received ataluren as oral powder for suspension at the dosages of 10, 10, and 20-mg/kg at morning, midday and evening, respectively for 48 weeks of treatment duration or until treatment discontinuation.
Period: Overall Study
Arm/Group | Ataluren | Placebo
Started | 140 | 139
Completed | 127 | 125
Not Completed | 13 | 14
Not completed — Withdrawal by Subject | 4 | 6
Not completed — Adverse Event | 3 | 4
Not completed — Physician Decision | 0 | 1
Not completed — Other Unspecified | 2 | 3
Not completed — Protocol Violation | 4 | 0

BASELINE CHARACTERISTICS:
Population: The as-treated population included all randomized participants who actually received any study treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Ataluren | Placebo | Total
Number analyzed (Participants) | 140 | 139 | 279
Age, Continuous [Mean (Standard Deviation); unit: years] | 22.0 (11.0) | 22.0 (10.44) | 22.0 (10.70)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 59 | 74 | 133
  Male | 81 | 65 | 146

OUTCOME MEASURES:

1. Primary Outcome: Absolute Change From Baseline in Percent-predicted Forced Expiratory Volume in One Second (ppFEV1) at Week 48
Description: The FEV1 is the volume of air forcibly exhaled in one second and is measured using forced expiratory air spirometry. Change in ppFEV1 at Week 48 was defined as the average between the change from baseline at Week 40 and that at Week 48. Baseline for ppFEV1 was defined as an average of ppFEV1 at Screening (Weeks -4 to -1) and Baseline (Day 1) visits.
Time Frame: From Baseline to Week 48
Population: The intent-to-treat (ITT) population included all randomized participants who had FEV1 data available at Baseline and at least one post-baseline visit.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage of predicted FEV1
Arm/Group | Ataluren | Placebo
Number analyzed (Participants) | 138 | 136
Percentage of predicted FEV1 | -1.396 [-2.7735 to -0.0180] | -1.992 [-3.3271 to -0.6576]
Statistical Analysis 1: Comparison: Ataluren vs Placebo; Test type: Superiority; p = 0.5336, Mixed-model, repeated-measures; Mean Difference (Net) = 0.597, 95% CI 2-sided [-1.2881 to 2.4813], Standard Error of Mean 0.9570

2. Secondary Outcome: 48-week Rate of Pulmonary Exacerbations
Description: Pulmonary exacerbations were assessed using expanded Fuchs criteria. The expanded Fuchs exacerbation is defined as the presence of at least 4 of 12 Fuchs' signs and symptoms requiring treatment with any form of antibiotic treatment (inhaled, oral, or intravenous). Fuchs' signs and symptoms included increased cough; change in sputum volume, color, or consistency; new or increased hemoptysis; increased dyspnea during moderate or mild exertion, or at rest; sinus pain or tenderness; change in sinus discharge; malaise, fatigue, or lethargy; anorexia or weight loss; temperature above 38 degrees Celsius; change in findings on chest examination; relative 10% decrease in ppFEV1, and chest radiography results consistent with pulmonary infection. The 48-week rate was calculated as: 48-week rate = total number of events /treatment duration by week*48.
Time Frame: Week 48
Population: The ITT population included all randomized participants who had FEV1 data available at Baseline and at least one post-baseline visit.
Measure: Mean (Standard Deviation); unit: number of exacerbations per 48 weeks
Arm/Group | Ataluren | Placebo
Number analyzed (Participants) | 138 | 136
number of exacerbations per 48 weeks | 0.950 (1.4038) | 1.127 (2.5241)
Statistical Analysis 1: Comparison: Ataluren vs Placebo; Test type: Superiority; p = 0.4008, Negative binomial regression; Rate ratio = 0.8567, 95% CI 2-sided [0.5973 to 1.2288], Standard Error of Mean 0.1577

3. Secondary Outcome: Change From Baseline in the Cystic Fibrosis Questionnaire - Revised (CFQ-R) Respiratory Domain at Week 48
Description: The teen/adult CFQ-R was used for this study. It was developed specifically for participants with cystic fibrosis. It is a disease-specific instrument designed to measure impact on overall health, daily life, perceived well-being, and symptoms. The respiratory domain assessed respiratory symptoms like coughing, congestion, wheezing etc. Scaling of each item is done via 4-point Likert scales. Scores for each item are summed up to generate a domain score. Scores ranges from 0 to 100, with higher scores indicating better health and lower scores indicating worse health.
Time Frame: Baseline (Day 1) and Week 48
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Ataluren | Placebo
Number analyzed (Participants) | 138 | 136
units on a scale | -0.760 [-3.4566 to 1.9364] | -1.032 [-3.7368 to 1.6728]
Statistical Analysis 1: Comparison: Ataluren vs Placebo; Test type: Superiority; p = 0.8881, Mixed-model, repeated measures; Mean Difference (Net) = 0.272, 95% CI 2-sided [-3.5292 to 4.0731], Standard Error of Mean 1.9300

4. Secondary Outcome: Change From Baseline in Body Mass Index (BMI) at Week 48
Description: Malnutrition is common in participants with cystic fibrosis. The BMI is an important clinical measure of nutritional status.
Time Frame: Baseline (Day 1) and Week 48
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: kilogram per meter square (kg/m^2)
Arm/Group | Ataluren | Placebo
Number analyzed (Participants) | 138 | 136
kilogram per meter square (kg/m^2) | 0.296 [0.1126 to 0.4789] | 0.361 [0.1759 to 0.5455]
Statistical Analysis 1: Comparison: Ataluren vs Placebo; Test type: Superiority; p = 0.6208, Mixed-model, repeated measures; Mean Difference (Net) = -0.065, 95% CI 2-sided [-0.3233 to 0.1934], Standard Error of Mean 0.1312

5. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs) and Treatment Emergent Serious Adverse Events (SAEs)
Description: An adverse event (AE) is any unfavourable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a study treatment, whether or not considered related to the study treatment. A TEAE is defined as an AE that occurs or worsens in the period extending from first dose of study drug to 4 weeks after last dose of study drug. An SAE is an untoward medical occurrence or effect associated with the use of a study drug at any dose, regardless of whether it is considered to be related to the study drug, which results in one of the following: death; inpatient hospitalization or prolongation of existing hospitalization; life threatening adverse event; persistent or significant disability or incapacity or substantial disruption of the ability to conduct normal life functions; any other medically important event; or a pregnancy resulting in spontaneous abortion, stillbirth, neonatal death, or congenital anomaly.
Time Frame: From study drug administration to 4-week post treatment follow-up visit (approximately 52 weeks)
Population: The as-treated population included all randomized participants who actually received any study treatment.
Measure: Number; unit: participants
Arm/Group | Ataluren | Placebo
Number analyzed (Participants) | 140 | 139
participants
  TEAEs | 133 | 135
  SAEs | 40 | 46

6. Secondary Outcome: Number of Participants With TEAEs by Severity and Relationship to Study Drugs
Description: The relationship of TEAEs to the study drugs were assessed as: probable related, possibly related, unlikely related, and unrelated. The severity of TEAEs were graded using the Common Terminology Criteria for Adverse Events, Version 3.0 as: Grade 1 (mild), Grade 2 (moderate), Grade 3 (severe), Grade 4 (life threatening), or Grade 5 (fatal).
Time Frame: From study drug administration to 4-week post treatment follow-up visit (approximately 52 weeks)
Population: The as-treated population included all randomized participants who actually received any study treatment.
Measure: Number; unit: participants
Arm/Group | Ataluren | Placebo
Number analyzed (Participants) | 140 | 139
participants
  Severity: Grade 1 | 26 | 18
  Severity: Grade 2 | 88 | 88
  Severity: Grade 3 | 19 | 29
  Severity: Grade 4 | 0 | 0
  Severity: Grade 5 | 0 | 0
  Relationship to study drug: Unrelated | 74 | 72
  Relationship to study drug: Unlikely related | 37 | 34
  Relationship to study drug: Possible related | 21 | 25
  Relationship to study drug: Probable related | 1 | 4

7. Secondary Outcome: Number of Participants With SAEs by Severity and Relationship to Study Drugs
Description: The relationship of SAEs to the study drugs were assessed as: probable related, possibly related, unlikely related, and unrelated. The severity of SAEs were graded using the Common Terminology Criteria for Adverse Events, Version 3.0 as: Grade 1 (mild), Grade 2 (moderate), Grade 3 (severe), Grade 4 (life threatening), or Grade 5 (fatal).
Time Frame: From study drug administration to 4-week post treatment follow-up visit (approximately 52 weeks)
Population: The as-treated population included all randomized participants who actually received any study treatment.
Measure: Number; unit: participants
Arm/Group | Ataluren | Placebo
Number analyzed (Participants) | 140 | 139
participants
  Severity: Grade 1 | 2 | 1
  Severity: Grade 2 | 23 | 20
  Severity: Grade 3 | 15 | 25
  Severity: Grade 4 | 0 | 0
  Severity: Grade 5 | 0 | 0
  Relationship to study drug: Unrelated | 26 | 31
  Relationship to study drug: Unlikely related | 13 | 15
  Relationship to study drug: Possible related | 1 | 0
  Relationship to study drug: Probable related | 0 | 0

8. Secondary Outcome: Number of Participants With Abnormal Vital Signs Reported as TEAEs
Description: Vital signs included systolic and diastolic blood pressure, pulse rate, pulse oximetry, and body temperature. Participants with abnormal vital signs who required clinical intervention or further investigation (beyond ordering a repeat [confirmatory] test) unless they are associated with an already reported clinical event are reported.
Time Frame: From study drug administration to 4-week post treatment follow-up visit (approximately 52 weeks)
Population: The as-treated population included all randomized participants who actually received any study treatment.
Measure: Number; unit: participants
Arm/Group | Ataluren | Placebo
Number analyzed (Participants) | 140 | 139
participants | 0 | 1

9. Secondary Outcome: Number of Participants With Abnormal Clinical Laboratory Parameters Reported as TEAEs
Description: Clinical laboratory tests included haematology, biochemistry, and urinalysis. Participants with abnormal laboratory parameters who required clinical intervention or further investigation (beyond ordering a repeat [confirmatory] test) unless they are associated with an already reported clinical event are reported.
Time Frame: From study drug administration to 4-week post treatment follow-up visit (approximately 52 weeks)
Population: The as-treated population included all randomized participants who actually received any study treatment.
Measure: Number; unit: participants
Arm/Group | Ataluren | Placebo
Number analyzed (Participants) | 140 | 139
participants | 32 | 30

10. Secondary Outcome: Number of Participants With Abnormal Electrocardiogram Reported as TEAEs
Description: Participants with abnormal electrocardiogram who required clinical intervention or further investigation (beyond ordering a repeat [confirmatory] test) unless they are associated with an already reported clinical event are reported.
Time Frame: From study drug administration to 4-week post treatment follow-up visit (approximately 52 weeks)
Population: The as-treated population included all randomized participants who actually received any study treatment.
Measure: Number; unit: participants
Arm/Group | Ataluren | Placebo
Number analyzed (Participants) | 140 | 139
participants | 1 | 0

ADVERSE EVENTS:
Time Frame: From study drug administration to 4-week post treatment follow-up visit (approximately 52 Weeks)
Description: All randomized participants who actually received any study treatment were analysed for AEs and SAEs.
Arm/Group | Ataluren | Placebo
All-Cause Mortality (participants affected / at risk) | 0/140 | 0/139
Serious Adverse Events (participants affected / at risk) | 40/140 | 46/139
Other Adverse Events (participants affected / at risk) | 123/140 | 120/139
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ataluren (N=140) | Placebo (N=139)
Infective pulmonary exacerbation of cystic fibrosis (Infections and infestations) | 25 (36) | 34 (50)
Pseudomonas infection (Infections and infestations) | 2 (2) | 0 (0)
Aspergillus infection (Infections and infestations) | 1 (1) | 0 (0)
Bronchopneumonia (Infections and infestations) | 1 (1) | 1 (2)
Bronchopulmonary aspergillosis allergic (Infections and infestations) | 1 (1) | 0 (0)
Device related sepsis (Infections and infestations) | 1 (1) | 0 (0)
Peritonitis (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 2 (2)
Pneumonia influenzal (Infections and infestations) | 1 (1) | 0 (0)
Respiratory tract infection (Infections and infestations) | 1 (2) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1)
Mycobacterium abscessus infection (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia staphylococcal (Infections and infestations) | 0 (0) | 1 (1)
Respiratory tract infection fungal (Infections and infestations) | 0 (0) | 1 (1)
Respiratory tract infection viral (Infections and infestations) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 0 (0) | 2 (2)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 1 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Nasal polyps (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Bronchopneumopathy (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumothorax spontaneous (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Distal intestinal obstruction syndrome (Gastrointestinal disorders) | 1 (1) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 3 (3) | 0 (0)
Renal failure acute (Renal and urinary disorders) | 1 (1) | 0 (0)
Pulmonary function test decreased (Investigations) | 1 (3) | 0 (0)
Forced expiratory volume decreased (Investigations) | 0 (0) | 1 (1)
Diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Red man syndrome (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Pseudocholinesterase deficiency (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Thrombosis in device (General disorders) | 0 (0) | 1 (1)
Costochondritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ataluren (N=140) | Placebo (N=139)
Diarrhoea (Gastrointestinal disorders) | 13 (15) | 12 (20)
Nausea (Gastrointestinal disorders) | 11 (14) | 10 (12)
Abdominal pain (Gastrointestinal disorders) | 11 (15) | 5 (6)
Vomiting (Gastrointestinal disorders) | 8 (8) | 4 (7)
Pyrexia (General disorders) | 9 (17) | 10 (12)
Infective pulmonary exacerbation of cystic fibrosis (Infections and infestations) | 75 (142) | 78 (145)
Viral upper respiratory tract infection (Infections and infestations) | 27 (43) | 21 (25)
Upper respiratory tract infection (Infections and infestations) | 21 (25) | 21 (26)
Sinusitis (Infections and infestations) | 16 (20) | 11 (11)
Nasopharyngitis (Infections and infestations) | 10 (13) | 8 (10)
Rhinitis (Infections and infestations) | 10 (12) | 8 (9)
Influenza (Infections and infestations) | 7 (7) | 8 (9)
Pharyngitis (Infections and infestations) | 7 (8) | 2 (3)
Pseudomonas infection (Infections and infestations) | 4 (4) | 9 (10)
Staphylococcal infection (Infections and infestations) | 4 (4) | 8 (9)
Back pain (Musculoskeletal and connective tissue disorders) | 7 (7) | 3 (7)
Headache (Nervous system disorders) | 12 (23) | 16 (18)
Cough (Respiratory, thoracic and mediastinal disorders) | 25 (36) | 25 (31)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 12 (17) | 10 (22)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No